CLINICAL TRIAL: NCT04231461
Title: Quality of Life After Cardiac Surgery
Acronym: QUACS
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: P02500
Record Dates: First submitted 2019-09-12; First posted 2020-01-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Stenosis; Mitral Valve Disease; Tricuspid Valve Disease; Aorta Disease; Coronary Artery Bypass Graft
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Cardiac Surgery — Routine or urgent cardiac surgery
  Other Names: Aortic Valve Procedure; Mitral Valve Procedure; Tricuspid Valve Procedure; Procedure on Aorta; Other major cardiac intervention; Other minimal access incisions

SUMMARY:
During the last twenty years heart surgery has become safer and the number of patients having heart surgery has increased with more frail patients being offered increasingly complex surgery. Heart operations often improve survival and quality of life (QoL), but that is not true for all patients. Regarding survival, clinicians can measure the risk to life from having a heart operation and the risk to life from not quite precisely, but clinicians have little idea about the impact of heart operations on QoL, which is the outcome that patients care about most. Clinicians are unable to provide patients with robust information on how an operation will affect their QoL. This study will provide this information by analysing the data from patient questionnaires immediately before and after the procedure and monthly thereafter for 12 months.

DETAILED DESCRIPTION:
The Sponsor shall use existing questionnaires to measure QoL in patients having major heart surgery. QoL will be measured before the operation and monthly afterwards for 12 months in order to answer the following questions:

1. How does having heart surgery affect the QoL immediately after the operation?
2. How long does it take patients to return to the same quality of life they had before the surgery?
3. How long does it take patients to regain any loss of quality of life due to the operation? Does quality of life improve thereafter?
4. What proportion of patients will achieve a net benefit in QoL?
5. Are there features that can predict who will benefit in terms of QoL and who will not? The Sponsor will use the data to develop an electronic calculator to enable quick and robust evaluation of the impact of heart surgery on the QoL of individuals. Patients will then be able to give truly informed consent and to decide if they wish have surgery based on a full knowledge of both surgical risk and the potential impact on QoL.

ELIGIBILITY:
Inclusion Criteria:

* EuroSCORE II ≥ 3% or EuroSCORE logistic of ≥ 6%
* Patients undergoing routine/ urgent cardiac surgery
* Patients must have the ability to provide informed consent

Exclusion Criteria:

* Patients undergoing salvage or emergency operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults able to understand the patient information sheet written in English.
Sampling Method: Non-Probability Sample
Enrollment: 2925 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life using Questionnaire EQ-5D | 12 Months
  Conduct questionnaire EQ-5D to assess Quality of Life Change post major cardiac surgery procedure. These questionnaires ask patients to assess their levels of pain, mobility, anxiety and depression to give an overall Quality of Life Measure.

SECONDARY OUTCOMES:
Change in Quality of Life using Questionnaire SF-12 | 12 Months
  Conduct questionnaire SF-12 to assess Quality of Life Change post major cardiac surgery procedure. These questionnaires ask patients to assess their levels of pain, mobility, anxiety and depression to give an overall Quality of Life Measure.

OTHER OUTCOMES:
Change in Quality of Life using Questionnaire LOT | 12 months
  Conduct questionnaire LOT to assess Quality of Life Change post major cardiac surgery procedure. These questionnaires ask patients to assess their levels of pain, mobility, anxiety and depression to give an overall Quality of Life Measure.
Change in Quality of Life using Questionnaire PANAS | 12 months
  Conduct questionnaire PANAS to assess Quality of Life Change post major cardiac surgery procedure. These questionnaires ask patients to assess their levels of pain, mobility, anxiety and depression to give an overall Quality of Life Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Samer Nashef, Study Director — Chief Investigator Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data is not to be shared with researchers